CLINICAL TRIAL: NCT07366684
Title: Investigation of Clinical Characteristics, Frailty, and Predictors of In-Hospital and Six-Month Prognosis in Hospitalized Patients Aged 75 Years and Older With Acute Coronary Syndrome
Brief Title: Clinical Characteristics, Frailty, and Prognostic Predictors in Patients Aged 75 and Older With Acute Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Clinical Center Niš (Other)
Collaborators: University of Nis (Other)
Responsible Party: Principal Investigator, Svetlana Apostolović, Full Professor of Internal Medicine, Head of the Department of Internal Medicine, Faculty of Medicine, University of Niš; Cardiologist at the Institute for Cardiology, Clinical Center Niš, Clinical Center Niš
Other Study IDs: ACS75-NIS-2025
Record Dates: First submitted 2025-12-01; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction; Non ST Elevation Myocardial Infarction (NSTEMI); Unstable Angina Pectoris
Keywords: Acute Coronary Syndrome (ACS); Elderly; Frailty; Percutaneous Coronary Intervention (PCI); Conservative Treatment; Major adverse cardiovascular events (MACE); Prognostic Predictors / Risk Stratification
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Acute Coronary Syndrome; Frailty | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized Patients ≥75 Years With Acute Coronary Syndrome: Patients aged 75 years and older admitted with acute coronary syndrome (STEMI, NSTEMI, or unstable angina). Data will be collected retrospectively and prospectively, including clinical, laboratory, echocardiographic, angiographic, and frailty parameters. Outcomes will be assessed during hospitalization and at 6 months after discharge.
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI); Other: Conservative Medical Therapy

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) — Patients receiving PCI as part of routine clinical care
Other: Conservative Medical Therapy — Patients treated conservatively with guideline-directed medical therapy as part of routine care

SUMMARY:
This study will evaluate clinical characteristics, frailty, and predictors of prognosis in patients aged 75 years and older who are hospitalized with acute coronary syndrome (ACS). The research includes both a retrospective and a prospective cohort. The aim is to determine whether frailty scores, combined with clinical and laboratory parameters available at admission, can improve risk prediction for complications and mortality compared with standard risk scores (TIMI, GRACE, Syntax). The study will also compare outcomes between patients treated with percutaneous coronary intervention (PCI) and those treated conservatively with medications. Patients will be followed during hospitalization and for six months after discharge. The results are expected to contribute to more personalized treatment strategies for elderly patients with ACS.

DETAILED DESCRIPTION:
This observational study will evaluate clinical characteristics,frailty, and prognostic predictors in patients aged 75 years and older hospitalized with acute coronary syndrome (ACS). The study is designed with two complementary components:

Retrospective cohort (≈350 patients):

Data will be collected from electronic medical records of patients previously hospitalized with ACS. Variables include demographics, comorbidities, laboratory findings (hematology, biochemistry, cardiac biomarkers), ECG changes, echocardiographic parameters, and coronary angiography results. Standard risk scores (TIMI, GRACE, Syntax) will be compared with observed outcomes. Data integrity will be ensured through double-entry verification, and missing values will be addressed using multiple imputation.

Prospective cohort (≈800 patients):

Patients will be consecutively enrolled at admission with ACS. Data collection will include the same parameters as in the retrospective cohort, with additional dynamic laboratory monitoring and frailty assesment. Frailty will be assessed within 48 hours of admission using the Rockwood Frailty Scale, performed by trained investigators. Echocardiography and coronary angiography will be conducted according to institutional protocols. Patients will be followed during hospitalization and 6 months after discharge, using structured case report forms and telephone interviews. Outcomes will include major adverse cardiovascular events (MACE), all-cause mortality, rehospitalizations, PCI-related complications (vascular, gastrointestinal bleeding, neurological), and treatment adherence.

Data management and statistical analysis:

All data will be entered into a secure, password-protected database with regular quality control checks. Statistical analyses will be performed using SPSS v.27 and R. Methods include descriptive statistics, univariate and multivariate logistic regression, ROC curve analysis, and comparison of AUC values. Predictors identified in the retrospective cohort will be validated in the prospective cohort.

The study team consists of cardiologists, statisticians, and trained research staff responsible for patient enrollment, frailty assessment, and data monitoring. Complications and adverse events will be defined according to standardized cardiology guidelines and adjudicated by an independent committee.

The study is conducted in accordance with the Declaration of Helsinki. Retrospective data collection does not require informed consent, while prospective participants will provide written informed consent. The expected contribution is improved risk stratification and more personalized therapeutic approaches for elderly patients with ACS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Diagnosis of acute coronary syndrome (STEMI, NSTEMI, or unstable angina)
* Hospitalization in a tertiary care center (University Clinical Center Niš)
* For prospective cohort: signed informed consent

Exclusion Criteria:

* Refusal to provide informed consent (prospective cohort)
* Missing or incomplete medical documentation (retrospective cohort)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients aged 75 years and older with acute coronary syndrome (STEMI, NSTEMI, unstable angina) treated at the University Clinical Center Niš. Approximately 350 retrospective and 200 prospective patients are expected to be included.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Impact of treatment strategy (PCI vs conservative therapy) on on all-cause mortality and major adverse cardiovascular events (MACE: cardiovascular death, myocardial infarction, stroke) in elderly patients with acute coronary syndrome (ACS) | Peri-procedurally (within 48 hours of PCI or index admission for conservative therapy), at discharge (assessed up to 14 days after admission (Day 1)), and at 6 months after discharge (± 14 days).
  To compare outcomes of patients aged ≥75 years with ACS (STEMI, NSTEMI, unstable angina) treated with percutaneous coronary intervention (PCI) versus conservative medical therapy. The primary outcome includes all-cause mortality and major adverse cardiovascular events (MACE). Unit of Measure: % of patients experiencing event.

SECONDARY OUTCOMES:
Impact of treatment strategy (PCI vs conservative therapy) on hemorrhagic complications | Peri-procedurally (within 48 hours of PCI or index admission) and at discharge (assessed up to 14 days after admission (Day 1)).
  Incidence of major bleeding, defined as clinically overt bleeding resulting in hemodynamic compromise, intracranial hemorrhage, bleeding requiring transfusion, or bleeding requiring surgical or endovascular hemostatic intervention; includes gastrointestinal and access-site bleeding. Unit of Measure: Incidence (%)
Number of Participants with ≥1 All-cause Rehospitalization | 6 months after discharge (± 14 days).
  Proportion of patients with ≥1 rehospitalization for any cause and total number of rehospitalizations per patient during follow-up; comparison between PCI and conservative therapy. Unit of Measure: % of patients with ≥1 rehospitalization; count per patient.
Demographic predictors of conservative management | Baseline (Day 1).
  Patient age and sex as predictors of the decision to pursue conservative medical therapy instead of percutaneous coronary intervention (PCI). Independent predictors will be identified using multivariable logistic regression and reported as odds ratios with 95% confidence intervals.
  Measure: Age (years); Sex (male/female).
Admission hemoglobin as predictor of conservative management | Baseline.
  Hemoglobin concentration measured at admission and recorded in the dataset. Evaluated as a predictor of conservative therapy versus PCI using multivariable logistic regression. Unit of Measure: g/L.
Admission eGFR (CKD-EPI) as predictor of conservative management | Baseline.
  Estimated glomerular filtration rate (CKD-EPI) measured at admission and recorded in the dataset. Evaluated as a predictor of conservative therapy versus PCI using multivariable logistic regression. Unit of Measure: mL/min/1.73 m².
Admission hs-Troponin I as predictor of conservative management | Baseline.
  High-sensitivity troponin I measured at admission; assay name and 99th percentile documented. Evaluated as a predictor of conservative therapy versus PCI using multivariable logistic regression. Unit of Measure: ng/L.
Admission CRP as predictor of conservative management | Baseline.
  C-reactive protein measured at admission and recorded in the dataset. Evaluated as a predictor of conservative therapy versus PCI using multivariable logistic regression. Unit of Measure: mg/L.
Admission BNP/NT-proBNP as predictor of conservative management | Baseline.
  BNP or NT-proBNP measured at admission and recorded in the dataset. Evaluated as a predictor of conservative therapy versus PCI using multivariable logistic regression. Unit of Measure: pg/mL.
Admission HbA1c as predictor of conservative management | Baseline.
  Glycated hemoglobin (HbA1c) measured at admission and recorded in the dataset. Evaluated as a predictor of conservative therapy versus PCI using multivariable logistic regression. Unit of Measure: %.
Composite admission laboratory abnormality score as predictor of conservative management | Baseline.
  Composite score derived from admission laboratory parameters not otherwise specified as individual outcomes. Included analytes: WBC with differential, RBC, HCT, MCV, MCH, MCHC, PLT, Glucose, urea, creatinine, total proteins, albumin, Total cholesterol, HDL, LDL, triglycerides, Na, K, Cl, Ca, AST, ALT, GGT, LDH, CK-MB, TSH.
  Each analyte will be coded as 1 if outside the central hospital laboratory reference range and 0 if within range (assay name, manufacturer, units, and reference intervals documented). The composite score equals the total number of abnormal parameters per patient and will be entered as a single predictor variable in multivariable logistic regression to evaluate its association with the decision for conservative therapy versus PCI. Missing data will be handled by multiple imputation; sensitivity analyses will assess robustness. Unit of Measure: Count (number of abnormal parameters per patient).
ECG ischemic changes at admission as predictor of conservative management | Baseline
  Binary composite coded as 1 if any of the following are present on the admission ECG: ST elevation, ST depression, T-wave inversion, or pathologic q/Q/qS complexes; coded as 0 if none are present. Evaluated as a predictor of conservative therapy versus PCI in multivariable logistic regression. Unit of measure: Presence/absence (yes/no).
ECG rhythm and arrhythmias at admission as predictor of conservative management | Baseline.
  Binary composite coded as 1 if any of the following are present on the admission ECG: atrial fibrillation (any), atrial flutter, supraventricular tachycardia, premature atrial complexes, premature ventricular complexes, non-sustained VT, sustained VT, ventricular fibrillation, or accelerated idioventricular rhythm; coded as 0 if none are present. Evaluated as a predictor of the decision for conservative therapy versus PCI. Unit of measure: Presence/absence (yes/no).
ECG conduction abnormalities at admission as predictor of conservative management | Baseline
  Binary composite coded as 1 if any of the following are present on the admission ECG: sinoatrial block, sick sinus syndrome, atrioventricular block (any degree), right bundle branch block, left bundle branch block, left anterior hemiblock, or left posterior hemiblock; coded as 0 if none are present. Evaluated as a predictor of the decision for conservative therapy versus PCI.
Angiographic high-risk anatomy composite as predictor of conservative management | Peri-procedurally (immediately after angiography); values used are those available at or prior to the documented treatment decision (decision documented within 48 hours of admission).
  Binary composite coded as 1 if any of the following are present on coronary angiography prior to the treatment decision: left main coronary lesion (≥50% luminal stenosis), multivessel coronary disease (≥2 epicardial vessels with significant stenosis), bifurcation lesion, or ≥70% stenosis in any vessel; coded as 0 if none are present. Evaluated as a predictor of the decision to pursue conservative medical therapy versus PCI in multivariable logistic regression. Unit of measure: Presence/absence (yes/no).
Left Ventricular Ejection Fraction as predictor of conservative management | At admission (transthoracic echo within 72 hours of admission), values used are those available at or prior to the documented treatment decision.
  Categorical coded as 1 if LVEF ≤40%, coded as 2 if 41-49%, coded as 3 if ≥50%, based on Teichholz, Simpson biplane, or visual estimation if biplane unavailable. Evaluated as a predictor of conservative therapy versus PCI in multivariable logistic regression. Examinations will be performed using the GE Healthcare Vivid 6 ultrasound system (General Electric) in our central echocardiography laboratory, following standardized protocols.
E/e' ratio as predictor of conservative management | At admission (transthoracic echo within 72 hours of admission), values used are those available at or prior to the documented treatment decision.
  Binary composite coded as 1 if average E/e' ≥16, coded as 0 if <16. Evaluated as a predictor of conservative therapy versus PCI in multivariable logistic regression. Examinations will be performed using the GE Healthcare Vivid 6 ultrasound system (General Electric) in our central echocardiography laboratory, following standardized protocols.
Pericardial effusion as predictor of conservative management | At admission (transthoracic echo within 72 hours of admission), values used are those available at or prior to the documented treatment decision.
  Binary coded as 1 if effusion present, coded as 0 if absent. Evaluated as a predictor of conservative therapy versus PCI in multivariable logistic regression. Examinations will be performed using the GE Healthcare Vivid 6 ultrasound system (General Electric) in our central echocardiography laboratory, following standardized protocols.
Left Atrial Volume Index as predictor of conservative management | At admission (transthoracic echo within 72 hours of admission), values used are those available at or prior to the documented treatment decision.
  Categorical coded as 1 if LAVI ≥34 mL/m², coded as 0 if <34 mL/m². Evaluated as a predictor of conservative therapy versus PCI in multivariable logistic regression. Examinations will be performed using the GE Healthcare Vivid 6 ultrasound system (General Electric) in our central echocardiography laboratory, following standardized protocols.
Wall Motion Score Index as predictor of conservative management | At admission (transthoracic echo within 72 hours of admission), values used are those available at or prior to the documented treatment decision.
  Categorical coded as 1 if WMSI >1.0, coded as 0 if ≤1.0. Evaluated as a predictor of conservative therapy versus PCI in multivariable logistic regression. Examinations will be performed using the GE Healthcare Vivid 6 ultrasound system (General Electric) in our central echocardiography laboratory, following standardized protocols.
Valvular regurgitation as predictor of conservative management | At admission (transthoracic echo within 72 hours of admission), values used are those available at or prior to the documented treatment decision.
  Binary composite coded as 1 if any of the following are present: aortic regurgitation, mitral regurgitation, pulmonary regurgitation, or tricuspid regurgitation; coded as 0 if none are present. Evaluated as a predictor of conservative therapy versus PCI in multivariable logistic regression. Examinations will be performed using the GE Healthcare Vivid 6 ultrasound system (General Electric) in our central echocardiography laboratory, following standardized protocols.
Comorbidity predictors of conservative management | At admission (baseline, pre-intervention/decision).
  Presence of predefined comorbid conditions recorded at admission and used as predictors of the decision for conservative therapy versus PCI. Each comorbidity will be recorded using standard clinical definitions and ICD codes where available. Comorbidities will be coded as binary variables (yes/no); chronic kidney disease will be classified by KDIGO stage (CKD stage 1-5). Candidate comorbid predictors will be evaluated in univariate analyses and included in multivariable logistic regression based on clinical relevance and univariate p<0.10. Missing data will be handled by multiple imputation; sensitivity analyses will be performed.
Frailty predictors of conservative management | At admission (baseline, pre-intervention/decision).
  Frailty assessed at admission using the Rockwood Clinical Frailty Scale (CFS) and the Hopkins frailty instrument; assessor initials and assessment timing recorded. Scores modeled primarily as continuous and secondarily as prespecified categorical variables; inclusion in multivariable logistic regression guided by univariate screening and clinical relevance; missing data handled by multiple imputation. Measure: Rockwood CFS coded as: 0 (score 1-3); 1 (score 4-6); 2 (score 7-9). Hopkins frailty coded as: 0 (score 0); 1 (score 1-2); 2 (score 3-5). Raw Rockwood CFS (1-9) and raw Hopkins score (numeric) will be recorded.
Number of Participants with Major Adverse Cardiovascular Events (MACE) | Outcome assessed at discharge (up to 14 days after admission (Day 1)), and outcomes reassessed 6 months after discharge (± 14 days).
  Composite endpoint defined as cardiovascular death, myocardial infarction, or stroke. Participants will be coded as positive if any of these events occur, and negative if none occur. Unit of measure: Presence/absence (yes/no).
Number of Participants with Cardiovascular Rehospitalization | Outcome assessed at discharge (up to 14 days after admission (Day 1)), and outcomes reassessed 6 months after discharge (± 14 days).
  Presence/absence of rehospitalization due to cardiovascular causes (including acute coronary syndrome, heart failure, arrhythmia, stroke, or repeat revascularization). Unit of measure: Presence/absence (yes/no).
Number of Participants with All-cause Mortality | Outcome assessed at discharge (up to 14 days after admission (Day 1)), and outcomes reassessed 6 months after discharge (± 14 days).
  Presence/absence of death from any cause. Unit of measure: Presence/absence (yes/no).
Correlation between clinical predictors and clinical outcomes (in-hospital MACE and 6-month all-cause mortality) | Predictors measured at admission (baseline). In-hospital MACE assessed during hospitalization (up to 15 days after admission). Six-month all-cause mortality assessed 6 months after discharge (±14 days).
  The outcomes are in-hospital major adverse cardiovascular events (MACE: cardiovascular death, myocardial infarction, stroke) and all-cause mortality at 6 months. Each outcome will be reported separately. Candidate predictors include demographic characteristics, prespecified comorbidities, admission laboratory values (including renal function and eGFR), echocardiographic measures (e.g., LVEF, LV volumes, LAVI, TAPSE), ECG parameters (e.g., ST elevation/depression, T-wave inversion, rhythm abnormalities, conduction blocks), and angiographic findings (culprit vessel, multivessel disease, left main disease, percent stenosis). Independent predictors will be identified using multivariable logistic regression for in-hospital MACE and Cox proportional hazards models for 6-month mortality. Full variable definitions, units, assay names, and reference ranges are provided in the SAP.
Correlation between frailty scores and cognitive categories and clinical outcomes (in-hospital MACE and 6-month all-cause mortality). | Scores measured at admission, outcomes assessed at discharge (up to 14 days after admission), and outcomes reassessed 6 months after discharge (± 14 days).
  Frailty and cognition will be assessed at admission using the Rockwood Clinical Frailty Scale (CFS, range 1-9; higher = greater frailty), the Hopkins frailty instrument (range 0-5; higher = greater frailty), and the Mini-Mental State Examination (MMSE, range 0-30; higher = better cognition). Clinical outcomes are in-hospital MACE (composite of cardiovascular death, myocardial infarction, and stroke) and all-cause mortality at 6 months. Results will be reported by the prespecified score categories (CFS 1-3 / 4-6 / 7-9; Hopkins 0 / 1-2 / 3-5; MMSE <24 vs ≥24) and expressed as the percentage of patients with each outcome within categories. Statistical analysis will include correlation coefficients (Spearman or Pearson as appropriate) and multivariable models comparing categories (logistic regression for in-hospital MACE; Cox proportional hazards for 6-month mortality); reference groups, covariates and all cutoffs are specified in the SAP.
Secondary complications and adverse events | Peri-procedurally, at discharge (assessed up to 14 days after admission (Day 1)), and at 6 months after discharge (± 14 days).
  Incidence of periprocedural complications, gastrointestinal bleeding, neurological complications, and psychiatric disorders (e.g., psycho-organic syndrome).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Center Niš, Niš, Serbia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographics, clinical, laboratory, echocardiographic, angiographic, frailty scores, and outcomes, will be made available. A data dictionary will also be provided. Data will be shared with qualified researchers upon reasonable request, after publication of the main results, for up to 5 years. Access will require approval by the principal investigator and a signed data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available after publication of the main results and will remain accessible for 5 years.
Access Criteria: Access will be granted to qualified researchers affiliated with academic or healthcare institutions for non-commercial scientific purposes. Requests must include a research proposal and data use agreement.

REFERENCES:
- [Background] Narendren A, Whitehead N, Burrell LM, Yudi MB, Yeoh J, Jones N, Weinberg L, Miles LF, Lim HS, Clark DJ, Al-Fiadh A, Farouque O, Koshy AN. Management of Acute Coronary Syndromes in Older People: Comprehensive Review and Multidisciplinary Practice-Based Recommendations. J Clin Med. 2024 Jul 28;13(15):4416. doi: 10.3390/jcm13154416. PMID 39124683
- [Background] Morici N, De Servi S, De Luca L, Crimi G, Montalto C, De Rosa R, De Luca G, Rubboli A, Valgimigli M, Savonitto S. Management of acute coronary syndromes in older adults. Eur Heart J. 2022 Apr 19;43(16):1542-1553. doi: 10.1093/eurheartj/ehab391. PMID 34347065
- [Background] H Ratcovich, P Palm, J Faerch, L Bang, T Engstroem, H H Tilsted, L Holmvang, Prevalence and prognosis of frailty in patients >70 years old with acute coronary syndrome referred to invasive angiography. Eur Heart J Acute Cardiovasc Care. 2023;12(Suppl 1):zuad036.045. doi:10.1093/ehjacc/zuad036.045
- [Background] Szummer K, Montez-Rath ME, Alfredsson J, Erlinge D, Lindahl B, Hofmann R, Ravn-Fischer A, Svensson P, Jernberg T. Comparison Between Ticagrelor and Clopidogrel in Elderly Patients With an Acute Coronary Syndrome: Insights From the SWEDEHEART Registry. Circulation. 2020 Nov 3;142(18):1700-1708. doi: 10.1161/CIRCULATIONAHA.120.050645. Epub 2020 Sep 1. PMID 32867508
- [Background] Aranzulla TC, Radano I, Civera S, Musumeci G. Acute coronary syndrome in elderly and frail patients. European Society of Cardiology - Council for Cardiology Practice, CardioPractice. Published August 6, 2024. Available at: https://www.escardio.org/Councils/Council-for-Cardiology-Practice-%28CCP%29/Cardiopractice/acute-coronary-syndrome-in-elderly-and-frail-patients
- [Background] Damluji AA, Forman DE, Wang TY, Chikwe J, Kunadian V, Rich MW, Young BA, Page RL 2nd, DeVon HA, Alexander KP; American Heart Association Cardiovascular Disease in Older Populations Committee of the Council on Clinical Cardiology and Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Radiology and Intervention; and Council on Lifestyle and Cardiometabolic Health. Management of Acute Coronary Syndrome in the Older Adult Population: A Scientific Statement From the American Heart Association. Circulation. 2023 Jan 17;147(3):e32-e62. doi: 10.1161/CIR.0000000000001112. Epub 2022 Dec 12. PMID 36503287
- [Background] Rout A, Moumneh MB, Kalra K, Singh S, Garg A, Kunadian V, Biscaglia S, Alkhouli MA, Rymer JA, Batchelor WB, Nanna MG, Damluji AA. Invasive Versus Conservative Strategy in Older Adults >/=75 Years of Age With Non-ST-segment-Elevation Acute Coronary Syndrome: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2024 Nov 5;13(21):e036151. doi: 10.1161/JAHA.124.036151. Epub 2024 Nov 4. PMID 39494560